CLINICAL TRIAL: NCT01344317
Title: The Effect of Stimulating Substances on Brain Activity Measured by Amplitude-integrated EEG and Long-term Neurodevelopmental Outcome of Preterm Infants Born Below 30 Weeks of Gestation
Brief Title: The Effect of Stimulating Substances on Brain Activity of Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christine Czaba, Dr.med.univ., Medical University of Vienna
Other Study IDs: Nationalbankprojekt Nr.13660
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Apneas of Prematurity
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Caffeine group: Premature infants below 30 weeks of gestation who receive Caffeine treatment
- Caffeine and Doxapram group: Premature infants below 30 weeks of gestation who receive Caffeine and Doxapram treatment
- Group with no treatment: Premature infants below 30 weeks of gestation with no stimulating treatment

SUMMARY:
Introduction: Methylxanthines and doxapram have been widely used for the treatment of apneas of prematurity. Both substances have effects on the central nervous system. While there are data available concerning the use of caffeine (the methylxanthine used at our NICU) even proposing a positive effect on neurodevelopmental outcome of very preterm infants, there are data which suggest a negative effect of the central stimulants doxapram on longterm outcome in this group of infants. Nevertheless concerning both medications only few studies have been published and only scarce data are available concerning the effect of these medications on brain activity of very preterm infants until now.

The aim of this study: is the assessment of the effect of stimulating substances on brain activity of preterm infants born below 30 weeks of gestation and their longterm neurodevelopmental follow-up.

Methods: This study is a prospective study including preterm infants born below 30 weeks of gestational age. Brain activity is measured by one-channel amplitude-integrated EEG (aEEG). The first aEEG measurement is performed without caffeine and/or doxapram medication. At least one hour of brain activity is registrated. The second measurement is done at least 24 hours after the start of caffeine and/ or doxapram treatment.

The percentage of different background patterns, the occurrence and duration of sleep-wake-cycling, and the occurrence and duration of seizures is assessed and analysed. Neurodevelopmental outcome is assessed at one and two years of corrected age by assessment of the Bayley Scales of Infant Development II and standardized clinical neurological examination.

ELIGIBILITY:
Inclusion Criteria:

see above

Exclusion Criteria:

* intraventricular hemorrhage
* posthaemorrhagic hydrocephalus
* cerebral infection
* cerebral malformation

Ages: 23 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants born below a gestational age of 30 weeks
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2016-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Weninger, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (2):
- Austria (2):
  - Medical University of Vienna, Department of Pediatrics and Adolescent Medicine, Neonatology, Vienna, Vienna
  - Medical University of Vienna, Vienna, Vienna